CLINICAL TRIAL: NCT00101504
Title: Partnership Programs to Reduce Cardiovascular Disparities - Hypertension Education and Treatment (HEAT)
Brief Title: Hypertension Education and Treatment Partnership for Reducing Ethnic Differences in the Risk of Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1286; U01HL079378 (NIH); U01HL079458 (NIH)
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2006-04

CONDITIONS: Cardiovascular Diseases; Hypertension; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Diseases

SUMMARY:
The purpose of this study is to improve hypertension outcomes in racial and ethnic minorities.

DETAILED DESCRIPTION:
BACKGROUND:

While there has been great progress in reducing CVD morbidity and mortality in the U.S. over the past 40 years, some minority groups have not shared fully in this progress and continue to have lower life expectancy and higher CVD morbidity. On average, minorities have less access to medical care, receive less aggressive care and fewer diagnostic and therapeutic cardiac procedures, and adhere poorly to prescribed medical regimens. Thus, research to reduce health disparities by improving CVD outcomes in minorities offers potential for a substantial positive public heath impact. Academic medical centers and institutions capable of carrying out such research, however, often lack access to and the trust of minority patients. Minority patients often receive fragmented care because they lack access to regular medical care, present to emergency departments rather than primary care physicians for complications of an advanced chronic CVD condition, and are less likely to follow medical regimens. Minority communities often harbor distrust of clinical research. Minority patients report greater satisfaction when receiving care from minority providers and are reluctant to receive treatment outside their minority healthcare serving systems.

In general, minorities have high rates of hypertension, elevated cholesterol, cigarette smoking, obesity, metabolic syndrome, and diabetes, as well as other behavioral, environmental, and occupational risk factors for cardiovascular diseases, such as sleep problems - all elements that contribute to excess CVD morbidity and mortality. The causes of minority health disparities are complex and incompletely understood. Although evidence of genetic, biologic, and environmental factors is well documented, poor outcomes are also attributed to under-treatment. Such under-treatment may be due to limited access to health care or, in some cases, break-down of the medical system, or failure of the physician and/or patient to allow for optimal health care, even when access is not impaired. The complex interactions of behavior, socio-economic status (SES), culture, and ethnicity are important predictors of health outcomes and sources of health disparities. Despite efforts to elucidate genetic and environmental risk factors and to promote cardiovascular health in high-risk populations, trends in CVD outcomes suggest that CVD health disparities continue to widen.

The Partnerships Program to Reduce Cardiovascular Health Disparities involves collaboration between research-intensive medical centers (RIMCs) that have a track record of NIH-supported research and patient care and minority healthcare serving systems (MSSs) that lack a strong research program. Each Partnership Program will: a) design and carry out multiple interdisciplinary research projects that investigate complex biological, behavioral, and societal factors that contribute to CVD health disparities and facilitate clinical research within the MSS to improve CVD outcomes and reduce health disparities, and b) provide reciprocal educational and skills development programs so that investigators will be able to conduct research aimed at reducing cardiovascular disparities and thereby enhance research opportunities, enrich cultural sensitivity, and improve cardiovascular research capabilities at both institutions.

The Request for Applications for Partnership Programs to Reduce Cardiovascular Disparities was released in September 2003. The awards were made in September 2004.

DESIGN NARRATIVE:

The University of Mississippi Medical Center (the Research Intensive Medical Center) and Jackson-Hinds Comprehensive Health Center (the Minority Healthcare Serving System) will address cardiovascular health disparities among African Americans through establishment of its HEAT Partnership. HEAT is an acronym for Hypertension Education and Treatment. The HEAT Partnership is organized into four cores. The administrative core includes the principal investigators from both the RIMC and the MSS as well as the core directors and co-directors. Specific aims of the Research Core are to: (1) provide a series of workshops for healthcare providers that focus on assessment and treatment of hypertensive patients according to current guidelines; (2) enroll a sufficient number of patients with uncontrolled hypertension to participate in the study and encourage each of them to continue treatment throughout the duration of the intervention as a means of promoting lifetime hypertension control; (3) provide a program of patient education that includes (a) a series of workshops for the intervention participants that focus on the impact of hypertension, and the efficacy of proper diet and exercise in managing hypertension; (b) a patient advocate, who will serve as a liaison between patient and provider; and (c) a "health partner" from the patient's social circle of acquaintances who will help reinforce the workshop lessons in a participatory manner; and (4) compare the results of the intervention group and the control group, and determine the effectiveness of the intervention. Specific aims of the Education Core are to: (1) enhance cultural competency among healthcare providers and address its impact on health disparities among the nation's racial and ethnic minority populations; (2) explore issues of race, racism, and health disparities in research and medical care, particularly as they affect African Americans in Mississippi; and (3) provide career development training for new investigators capable of conducting research to reduce cardiovascular health disparities. Specific aims of the Community Outreach Core are to: (1) conduct focus group sessions in selected vulnerable populations to assess the level of awareness about hypertension and identify realistic lifestyle hypertension-prevention goals for the intended audience; (2) pursue partnerships with community-based organizations to enhance the activities of the Outreach Core; and (3) develop and disseminate culturally and linguistically appropriate education materials to the lay public about hypertension, including detection, diagnosis, and strategies for its prevention.

The study completion date listed in this record was obtained from the "End Date" entered in the Query View Report (QVR) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-09; Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Gordon, Principal Investigator — Jackson Hinds Comprehensive Health Center; Herman Taylor, Principal Investigator — University of Mississippi Medical Center